CLINICAL TRIAL: NCT00465569
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Oral Milk Immunotherapy for Cow's Milk Allergy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00002102
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Milk Hypersensitivity
Keywords: Food Allergy; Oral Immunotherapy; Immunoglobulin E
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Treatment (Experimental): Pre-measured doses of dry, nonfat powered milk prepared by the clinical research-registered dieticians
  Interventions: Drug: cow's milk powder
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: cow's milk powder — Milk powder given orally in escalating doses to a goal of 500 mg for approximately 23 weeks
  Arms: Active Treatment
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if small oral doses of milk protein are safe and effective in decreasing sensitivity to cow's milk in allergic children.

DETAILED DESCRIPTION:
This is a prospective, multi-center, clinical trial involving children aged 6 to 21 years with persistent cow's milk allergy. These children will be recruited from 2 sites (Johns Hopkins and Duke University) and will undergo initial screening and double-blind, placebo-controlled, food challenge (DBPCFC) to confirm threshold dose for reactivity to milk. Patients will be treated with milk oral immunotherapy (OIT) or placebo for 22-30 weeks. Those who reach an adequate maintenance dose for OIT will undergo a second DBPCFC. Those who develop desensitization will continue with daily milk intake and undergo a third DBPCFC. Those in the treatment group who are not desensitized will return to strict avoidance. Those in placebo group will be offered to begin treatment or continue with strict milk avoidance. Symptom and diet information will be collected initially and at regular intervals. Bloodwork, skin prick tests (SPTs), pulmonary function tests (PFTs), and oral secretion samples will be done initially and at periodic intervals.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent (by parent or legal guardian if the subject is a minor) and informed assent if applicable
* Age 6 to 21 years
* Must have history of symptomatic reactivity to cow's milk (eczema, urticaria, upper/lower resp., GI, other associated rash, oral symptoms)
* History of positive skin prick test (wheal >/= histamine control) or milk-Immunoglobulin E (IgE)>0.35 kilounits per liter (kU/L)
* Positive DBPCFC
* All females of child bearing age must be using appropriate birth control

Exclusion Criteria:

* History of anaphylaxis requiring hospitalization
* History of intubation related to asthma
* Has the ability to tolerate >2.4gram of milk protein at initial DBPCFC
* Has a history of allergy to any component of vehicle
* Pregnancy (need negative test)
* Viral upper respiratory infection (URI) or gastroenteritis within 7days of OFC (OFC needs to be rescheduled)
* Has pulmonary function tests <80% of predicted (FEV1) or clinical history consistent with moderate persistent asthma
* Currently taking greater than medium dose inhaled corticosteroid (>400mcg/day fluticasone or fluticasone equivalent if </=12yo or >600mcg/day if >12 years old)
* Antihistamine within 1 week prior to skin testing or food challenges (Skin testing and/or food challenge needs to be rescheduled)
* Systemic corticosteroid within 4 weeks prior to baseline visit
* Receiving omalizumab, beta-blocker, Angiotensin-converting enzyme (ACE) inhibitor or tricyclic antidepressant therapy
* Chronic disease (other than asthma, atopic dermatitis, rhinitis) requiring therapy (e.g., heart disease, diabetes)
* Participation in any interventional study for treatment of a food allergy in the past 12 months
* Severe reaction at initial DBPCFC, defined as:

  i. Life-threatening anaphylaxis ii. Requires overnight hospitalization

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Wood, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Duke University, Durham, North Carolina

REFERENCES:
- [Background] Buchanan AD, Green TD, Jones SM, Scurlock AM, Christie L, Althage KA, Steele PH, Pons L, Helm RM, Lee LA, Burks AW. Egg oral immunotherapy in nonanaphylactic children with egg allergy. J Allergy Clin Immunol. 2007 Jan;119(1):199-205. doi: 10.1016/j.jaci.2006.09.016. Epub 2006 Oct 27. PMID 17208602
- [Background] Meglio P, Bartone E, Plantamura M, Arabito E, Giampietro PG. A protocol for oral desensitization in children with IgE-mediated cow's milk allergy. Allergy. 2004 Sep;59(9):980-7. doi: 10.1111/j.1398-9995.2004.00542.x. PMID 15291907
- [Background] Enrique E, Pineda F, Malek T, Bartra J, Basagana M, Tella R, Castello JV, Alonso R, de Mateo JA, Cerda-Trias T, San Miguel-Moncin Mdel M, Monzon S, Garcia M, Palacios R, Cistero-Bahima A. Sublingual immunotherapy for hazelnut food allergy: a randomized, double-blind, placebo-controlled study with a standardized hazelnut extract. J Allergy Clin Immunol. 2005 Nov;116(5):1073-9. doi: 10.1016/j.jaci.2005.08.027. Epub 2005 Oct 3. PMID 16275379
- [Result] Skripak JM, Nash SD, Rowley H, Brereton NH, Oh S, Hamilton RG, Matsui EC, Burks AW, Wood RA. A randomized, double-blind, placebo-controlled study of milk oral immunotherapy for cow's milk allergy. J Allergy Clin Immunol. 2008 Dec;122(6):1154-60. doi: 10.1016/j.jaci.2008.09.030. Epub 2008 Oct 25. PMID 18951617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children between the ages of 6 and 21 years with a known history of IgE-mediated milk allergy were recruited from the pediatric allergy clinics at the Johns Hopkins University Hospital, Baltimore, Maryland, and Duke University Medical Center, Durham, North Carolina.
Pre-assignment Details: Eligibility criteria were a positive skin prick test (SPT) response to milk extract (wheal ≥ histamine control) or milk immunoglobulin E (IgE) level of > 0.35 kilounits per liter (kU/L) and a positive milk challenge result at baseline defined as reacting with clear signs, symptoms, or both to a cumulative dose of 2.5 g or less of milk protein.
Groups:
- Placebo: Pre-measured doses of ProFree, a dry, milk free powder
Period: Overall Study
Arm/Group | Active Treatment | Placebo
Started | 13 | 7
Completed | 12 | 7
Not Completed | 1 | 0
Not completed — persistent eczema during dose escalation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 7 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (3.3) | 10.2 (3.3) | 9.5 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20
History of eczema [Count of Participants; unit: Participants] | 7 | 4 | 11
Current eczema [Count of Participants; unit: Participants] | 4 | 2 | 6
History of asthma [Count of Participants; unit: Participants] | 12 | 5 | 17
Current asthma [Count of Participants; unit: Participants] | 9 | 3 | 12
History of other food allergy [Count of Participants; unit: Participants] | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: The Median Milk Threshold Dose Inducing a Reaction
Time Frame: Baseline and 23 weeks
Population: One participant in the active treatment arm did not complete the study due to persistent eczema during dose escalation. The median milk threshold dose in both groups was 40 with a full range of 40-1340 at the baseline challenge.
Measure: Median (Full Range); unit: miligrams
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 12 | 7
miligrams
  Baseline | 40 [40 to 1340] | 40 [40 to 1340]
  Change at 23 weeks | 5100 [2500 to 8100] | 0 [-1300 to 0]

2. Secondary Outcome: Changes in Cow Milk-IgE
Description: IgE is measured in kilounits per liter (kU/L). Measurements were obtained at Baseline and at 23 weeks
Time Frame: Baseline and 23 weeks
Population: One participant in the active treatment arm did not complete the study due to persistent eczema during dose escalation
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 12 | 7
percentage of change | 8 [-50 to 64] | -5 [-13 to 71]

3. Secondary Outcome: Changes in Cow Milk Immunoglobulin G4 (IgG4)
Description: IgG4 is measured in ug/mL. Measurements were obtained at Baseline and at 23 weeks
Time Frame: Baseline and 23 weeks
Population: One participant in the active treatment arm did not complete the study due to persistent eczema during dose escalation
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Active Treatment | Placebo
Number analyzed (Participants) | 12 | 7
percentage of change | 767 [29 to 1321] | 14 [-14 to 157]

ADVERSE EVENTS:
Groups:
- Active Treatment: Adverse event information is based on percentages of doses. There were 2437 total doses in the active treatment arm with a median of 177 and a range of 155-242 per participant. There was a total of 13 participants in the active treatment arm who were analyzed for the Adverse Events data reported below.
- Placebo: Adverse event information is based on percentages of doses. There were 1193 total doses in the placebo arm with a median of 171 and a range of 152-199 per participant. There was a total of 7 participants in the placebo arm who were analyzed for the Adverse Events data reported below.
Arm/Group | Active Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2437 | 0/1193
Serious Adverse Events (participants affected / at risk) | 0/2437 | 0/1193
Other Adverse Events (participants affected / at risk) | 1107/2437 | 134/1193
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=2437) | Placebo (N=1193)
Local symptoms (Skin and subcutaneous tissue disorders) | 870 (870) | 104 (104)
Gastrointestinal (Gastrointestinal disorders) | 458 (458) | 16 (16)
Lower respiratory (Respiratory, thoracic and mediastinal disorders) | 198 (198) | 28 (28)
Skin (Skin and subcutaneous tissue disorders) | 22 (22) | 1 (1)
Multiple systems (General disorders) | 29 (29) | 0 (0)
Eczema flare (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No